CLINICAL TRIAL: NCT04576975
Title: Perioperative Use of Ketamine Infusion vs Dexmedetomidine Infusion as Analgesic in Obese Patients Undergoing Bariatric Surgery
Brief Title: Ketamine Infusion vs Dexmedetomidine Infusion in Obese Patients Undergoing Bariatric Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Collaborators: Ministry of Health, Kuwait (Other Government)
Responsible Party: Principal Investigator, Belal Nabil Mahfouz Khalil, Assistant Lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU M D 108 / 2020
Record Dates: First submitted 2020-09-26; First posted 2020-10-06 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Morbid Obesity; Surgery
MeSH Terms: conditions — Obesity, Morbid | interventions — Ketamine; Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Blinding of patients and assigning them randomly to their groups will be done by giving patients serial numbers, using a computer program (Microsoft Excel 365). Investigators will be blinded to group assignments and drug coding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ketamine (Experimental): This group will receive a bolus dose of Ketamine [Ketamine HCL - Sterop, Belgium] (0.3 mg/kg) by the ideal body weight diluted with 0.9% Normal Saline over 10 minutes by 20 ml syringe infused before induction. After which Ketamine infusion (500 mg vial diluted over 50 cc infusion syringe, concentration 10 mg/ml) will start with rate of 0.3 mg/kg/hr till 10 Minutes before the end of the surgery
  Interventions: Drug: Ketamine
- Dexmedetomidine (Experimental): This group will receive a bolus dose of Dexmedetomidine [Precedex® -Hospira, USA] (0.5 µcg/kg) by the ideal body weight diluted with 0.9% Normal Saline over 10 minutes by 20 ml syringe infused before induction. After which, the Dexmedetomidine infusion (200 µcg vial diluted over 50 cc infusion syringe, concentration 4 µcg/ml) will start with rate of 0.5 µcg/kg/hr till 10 Minutes before the end of the surgery
  Interventions: Drug: Dexmedetomidine
- Normal Saline 0.9% (Placebo Comparator): This group will receive a bolus dose of NS 0.9% over 10 minutes by 20 ml syringe infused before induction. After which, NS 0.9% (50 ml over 50 cc syringe) will be infused.
  Interventions: Drug: Normal Saline 0.9%

INTERVENTIONS:
Drug: Ketamine — compare the use of ketamine versus dexmedetomidine when used as perioperative infusion in obese patients undergoing laparoscopic bariatric surgery regarding their analgesic efficacy as well as any side effects or drawbacks (PONV and effects on consciousness) that might associate with their use.
  Arms: Ketamine
Drug: Dexmedetomidine — compare the use of ketamine versus dexmedetomidine when used as perioperative infusion in obese patients undergoing laparoscopic bariatric surgery regarding their analgesic efficacy as well as any side effects or drawbacks (PONV and effects on consciousness) that might associate with their use.
  Arms: Dexmedetomidine
Drug: Normal Saline 0.9% — compare the use of ketamine versus dexmedetomidine when used as perioperative infusion in obese patients undergoing laparoscopic bariatric surgery regarding their analgesic efficacy as well as any side effects or drawbacks (PONV and effects on consciousness) that might associate with their use.
  Arms: Normal Saline 0.9%

SUMMARY:
The surgeries that involve treatment of morbid obesity, i.e. bypass procedure and sleeve gastrectomy, are collectively covered under the term 'bariatric surgery'. The frequency of bariatric surgery has been increasing worldwide for patients with medically complicated obesity who have difficulty losing weight by other methods

The growth of bariatric surgery is accompanied with development of anesthetic techniques to maintain patient safety and improve outcome. Treatment with narcotics in obese patients has dual effect. Increased use of narcotics are associated with multiple complications including Postoperative Nausea and Vomiting (PONV) , respiratory depression and elevated risk of Obstructive Sleep Apnea (OSA) complications . On the other hand, the reduction in opioid use may result in acute post-operative pain that may limit post-surgery rehabilitation. Therefore, we need to minimize opioid use and employ some other drugs which, besides having analgesia, has an opioid-sparing effect also.

Ketamine, an N-methyl-D-aspartate (NMDA) receptor antagonist, has analgesic properties in sub-anesthetic doses. When used in low dose (0.3 to 0.5 mg/kg) by ideal body weight, it is an analgesic, anti-hyperalgesic, and prevents development of opioid tolerance.

Dexmedetomidine is selective α2-Adrenoceptor agonist that has been used as an adjuvant to anesthetic agents in perioperative period for several adventitious profile as well as tolerated side effects . While dexmedetomidine is emerging as a beneficial adjunct to the analgesic regimen in the perioperative period, its utilization is not routinely widespread .

ELIGIBILITY:
Inclusion Criteria:

* BMI > 35 kg/m2
* ASA physical status II & III (according to BMI)
* Undergoing laparoscopic bariatric surgery

Exclusion Criteria:

* Patients refusal
* ASA physical status: IV (according to BMI)
* History of hypersensitivity to dexmedetomidine and/or ketamine
* History of substance abuse (Benzodiazepines) or Chronic opioid use
* Psychiatric or Seizure disorder
* uncontrolled hypertension or heart block
* uncontrolled diabetes
* Surgical Complication

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
compare the use of ketamine versus dexmedetomidine when used as perioperative infusion in obese patients undergoing laparoscopic bariatric surgery regarding their analgesic efficacy | one year throughout the study
  They will be assessed for sedation score with Modified Observer's assessment of alertness/sedation scale [MOAS/S] . The score will be repeated at 10, 30 and 60 minutes.
  Agitated 6 Responds readily to name spoken in normal tone (alert) 5 Lethargic response to name spoken in normal tone 4 Responds only after name is called loudly and/or repeatedly 3 Responds only after mild prodding or shaking 2 Does not respond to mild prodding or shaking 1 Does not respond to deep stimulus 0
  The patient will be assessed for pain by using the Numerical Rating Scale [NRS] with score is 0 for no pain and 10 for excruciating pain. The NRS score will be recorded 30 and 60 mins and 2, 6, 12, and 24 h after the surgery.
  All patients will receive paracetamol (Perfilgan ®) 1 gm IV every 6 hours for 24 hours postoperatively. A rescue dose of morphine 4 mg per needed with minimum 6 hours interval between doses if the NRS Score is ≥ 4. total doses of morphine will be calculated.

SECONDARY OUTCOMES:
any side effects or drawbacks (PONV and effects on consciousness) that might associate with their use | one year throughout the study
  All Patients will be assessed for PONV by using PONV Intensity Scale . The score will be done 6 hours and 24 hours after the surgery. Ondansetron (Zofran®) 4 mg will be given if the patient developed intense sensation of nausea and to be repeated after 30 Minutes
  All the vital data will be recorded at 10 minutes, 30 minutes, 1 hour, 2 hours, 6 hours, 12 hours and 24 hours from discharge of operating room.
  Postoperative complication (such as; airway obstruction, development of hypoxia, serious nausea and vomiting …, etc.) will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Bahaa El-Din E Ali, PhD, Study Director — Ainshams University, Egypt; Ahmed N El-Shaer, PhD, Study Director — Ainshams University, Egypt; Mohammad A Khaja, FCARCSI, Study Director — Ministry of Health, Kuwait; Mohammed O Taeimah, PhD, Principal Investigator — Ainshams University, Egypt; Maha S Al Derh, PhD, Principal Investigator — Ainshams University, Egypt; Belal N Khalil, M.Sc, Principal Investigator — Ainshams University, Egypt
Locations (1):
- Ainshams University Hospitals, Cairo, Egypt

REFERENCES:
- [Background] Albaugh VL, Abumrad NN. Surgical treatment of obesity. F1000Res. 2018 May 21;7:F1000 Faculty Rev-617. doi: 10.12688/f1000research.13515.1. eCollection 2018. PMID 29904577
- [Background] Hjermstad MJ, Fayers PM, Haugen DF, Caraceni A, Hanks GW, Loge JH, Fainsinger R, Aass N, Kaasa S; European Palliative Care Research Collaborative (EPCRC). Studies comparing Numerical Rating Scales, Verbal Rating Scales, and Visual Analogue Scales for assessment of pain intensity in adults: a systematic literature review. J Pain Symptom Manage. 2011 Jun;41(6):1073-93. doi: 10.1016/j.jpainsymman.2010.08.016. PMID 21621130
- [Background] Ingrande J, Lemmens HJ. Dose adjustment of anaesthetics in the morbidly obese. Br J Anaesth. 2010 Dec;105 Suppl 1:i16-23. doi: 10.1093/bja/aeq312. PMID 21148651
- [Background] Liu FL, Cherng YG, Chen SY, Su YH, Huang SY, Lo PH, Lee YY, Tam KW. Postoperative recovery after anesthesia in morbidly obese patients: a systematic review and meta-analysis of randomized controlled trials. Can J Anaesth. 2015 Aug;62(8):907-17. doi: 10.1007/s12630-015-0405-0. Epub 2015 May 22. PMID 26001751
- [Background] Nonaka T, Inamori M, Miyashita T, Inoh Y, Kanoshima K, Higurashi T, Ohkubo H, Iida H, Fujita K, Kusakabe A, Gotoh T, Nakajima A. Can sedation using a combination of propofol and dexmedetomidine enhance the satisfaction of the endoscopist in endoscopic submucosal dissection? Endosc Int Open. 2018 Jan;6(1):E3-E10. doi: 10.1055/s-0043-122228. Epub 2018 Jan 12. PMID 29340293
- [Background] Vaughns JD, Martin C, Nelson J, Nadler E, Quezado ZM. Dexmedetomidine as an adjuvant for perioperative pain management in adolescents undergoing bariatric surgery: An observational cohort study. J Pediatr Surg. 2017 Nov;52(11):1787-1790. doi: 10.1016/j.jpedsurg.2017.04.007. Epub 2017 Apr 19. PMID 28465076
- [Background] Wang J, Echevarria GC, Doan L, Ekasumara N, Calvino S, Chae F, Martinez E, Robinson E, Cuff G, Franco L, Muntyan I, Kurian M, Schwack BF, Bedrosian AS, Fielding GA, Ren-Fielding CJ. Effects of a single subanaesthetic dose of ketamine on pain and mood after laparoscopic bariatric surgery: A randomised double-blind placebo controlled study. Eur J Anaesthesiol. 2019 Jan;36(1):16-24. doi: 10.1097/EJA.0000000000000860. PMID 30095550
- [Background] Wengritzky R, Mettho T, Myles PS, Burke J, Kakos A. Development and validation of a postoperative nausea and vomiting intensity scale. Br J Anaesth. 2010 Feb;104(2):158-66. doi: 10.1093/bja/aep370. Epub 2009 Dec 26. PMID 20037151
- [Derived] Khalil BNM, Elderh MSH, Khaja MAR, El-Shaer AN, Ali BEEH, Taeimah MOA. Perioperative use of ketamine infusion versus dexmedetomidine infusion for analgesia in obese patients undergoing bariatric surgery: a double-blinded three-armed randomized controlled trial. BMC Anesthesiol. 2023 Apr 1;23(1):108. doi: 10.1186/s12871-023-02059-3. PMID 37005580